CLINICAL TRIAL: NCT00589290
Title: A Multicenter Phase II Study of Belinostat (PXD-101) in Previously Chemotherapy Treated Thymoma and Thymic Carcinoma
Brief Title: Belinostat (PXD101) to Treat Tumors of the Thymus at an Advanced Stage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080033; 08-C-0033; NCT00720187 (obsolete NCT alias)
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: Histone deacetylase (HDAC) Inhibitors; Mediastinal Neoplasm; Thymic Carcinoma; Thymoma
MeSH Terms: conditions — Thymoma; Mediastinal Neoplasms | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belinostat Treatment (Experimental): 1000 mg/m^2/day as a 30 minute intravenous (IV) infusion daily for 5 days every 3 weeks (day 1-5 of the 3 week treatment cycle). After 12 cycles of treatment, cycles will be given for 5 days every 4 weeks.
  Interventions: Drug: Belinostat (PDX101)

INTERVENTIONS:
Drug: Belinostat (PDX101) — 1000 mg/m^2/day as a 30 minute intravenous (IV) infusion daily for 5 days every 3 weeks (day 1-5 of the 3 week treatment cycle). After 12 cycles of treatment, cycles will be given for 5 days every 4 weeks.
  Other Names: PDX101

SUMMARY:
Background:

* Cisplatin-containing chemotherapy is the standard treatment for advanced tumors of the thymus that cannot be removed surgically.
* New treatment options are needed for patients with advanced tumors of the thymus that do not improve with cisplatin-containing therapy.
* Belinostat is a drug that inhibits enzymes called histone deacetylase. Histone deacetylase inhibitors have shown promising activity in many cancers and may be useful in treating patients with thymic tumors.

Objectives:

-To assess the safety and effectiveness of belinostat for treatment of malignant thymic tumors in patients who failed after standard treatment.

Eligibility:

-Patients 18 years of age or older with an advanced thymic tumor that has progressed after treatment with platinum-containing chemotherapy.

Design:

* Patients receive belinostat treatment in 21-day cycles. The drug is given as an infusion through a vein during days 1 through 5 of each cycle. Treatment cycles continue as long as the medicine is tolerated and the cancer does not worsen.
* Patients have a physical examination and several blood tests during every cycle.
* Patients have an electrocardiogram every cycle before starting the belinostat infusion and again on the last day of the infusion.
* Patients undergo computed tomography (CT) or other imaging test, such as ultrasound or MRI, every two cycles to evaluate the response of the tumor to treatment.
* Tumor tissue obtained from a previous biopsy is used for research purposes.

DETAILED DESCRIPTION:
Background:

Cisplatin-containing chemotherapy is the standard of care for advanced unresectable thymoma and thymic carcinoma. New options for treatment are necessary in patients with advanced thymoma and thymic carcinoma that have progressed on cisplatin-containing therapy. Histone deacetylase inhibitors have shown promising clinical activity in many malignancies. Belinostat, a potent histone deacetylase inhibitor, is a promising agent, which may have activity in patients with thymic malignancies.

Objectives:

* To assess objective response rate according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria for belinostat monotherapy.
* To assess safety of belinostat.
* To evaluate time to response, duration of response, progression-free survival and overall survival.
* To identify chromosomal gains or losses and gene methylation status by comparative genomic hybridization and methylation microarrays in thymoma / thymic carcinomas in relation to clinical outcome.
* To assess expression levels of particular proteins on the pretreatment tumor sample, by immunohistochemistry (IHC) and correlate them with clinical outcome.
* To identify and measure changes in p21 and protein hyperacetylation in peripheral blood mononuclear cells (PBMC), and vascular endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF) in plasma and correlate them with clinical outcome.
* To measure changes in modulation of T-cell function in peripheral blood lymphocytes.

Eligibility:

* Patients with histologically confirmed thymic carcinoma or thymoma who have previously been treated on at least one platinum containing chemotherapy regimen.
* Measurable disease by RECIST criteria.
* Adequate renal, hepatic and hematopoietic function.
* QT Interval must be less than 500 msec at baseline by electrocardiogram (EKG) (Fridericia's formula used for correction).
* No major surgery, radiotherapy, or chemotherapy within 28 days of belinostat therapy.

Design:

* Patients will receive belinostat as a 30-minute intravenous (IV) infusion of 1000 mg/m^2/day during days 1-5 every 3 weeks. After 12 cycles of treatment, cycles will be given every 4 weeks.
* Treatment with belinostat alone will continue until disease progression.
* Toxicity will be assessed every cycle by the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 until December 31, 2010, and by CTCAE Version 4.0 beginning January 1, 2011.
* Tumor response assessments by RECIST criteria will be performed every 2 cycles. After 12 cycles, response assessment will be every 3 cycles.
* Correlative studies including comparative genomic hybridization, methylation microarray analysis, and tissue immunohistochemistry studies will be done on existing tumor blocks.
* Blood samples for circulating plasma biomarkers of response including VEGF will be drawn the first day of cycle 1 and 2 as well as cycle 1, day 3.
* Blood samples for protein hyperacetylation and T cell modulation analyses will be drawn the first day of cycle 1 and 2.

ELIGIBILITY:
* INCLUSION CRITERIA:

Histologically confirmed invasive recurrent or metastatic thymoma or thymic carcinoma by the pathology department / Center for Cancer Research (CCR) / National Cancer Institute (NCI).

Patients must have had at least one prior platin-containing chemotherapy regimen. There is no limit to the number of prior chemotherapy regimens received. Progressive disease should have been documented before entry into the study.

Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as greater than 10 mm with spiral computed tomography (CT) scan.

Patients must have recovered from toxicity related to prior therapy to at least to grade 1 (defined by the Common Terminology Criteria for Adverse Events (CTCAE) 3.0 until December 31, 2010, and by CTCAE 4.0 beginning January 1, 2011) and must not have had prior chemotherapy within 4 weeks. Patients must be at least 28 days since any prior radiation or major surgery.

* Target lesions cannot be selected within previously irradiated areas, if not newly arising or clearly progressing after irradiation as proven by repeat scanning.
* Concurrent corticosteroids for myasthenia gravis, or other paraneoplastic syndromes, or other chronic conditions are allowed.

Age greater than 18 years.

Life expectancy of greater than 3 months.

Performance status (Eastern Cooperative Oncology Group (ECOG)) less than or equal to 2.

Patients must have adequate organ and marrow function (as defined below). Patients must have returned to base line or grade one from any acute toxicity related to prior therapy.

Laboratory Test/Required Value:

Absolute neutrophil count greater than 1,500/microl.

Platelets greater than 100,000/microl.

International normalized ratio (INR) less than or equal to 1.5 times upper limit of normal (ULN) or

Partial thromboplastin time (PTT) abnormality can be explained by the presences of lupus anticoagulant or in the therapeutic range if on anticoagulation.

Total bilirubin less than or equal to 1.5 times institutional upper limits of normal.

Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase(SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase(SGPT) less than or equal to 3 times institutional upper limit of normal.

Creatinine less than or equal to 1.5 times institutional upper limits of normal or Calculated Creatinine greater than 45 mL/min/1.73 m^2 for patients with creatinine.

Clearance levels above institutional normal.

The effects of belinostat on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because histone deacetylase (HDAC) inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and continue for at least 2 months after completion. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belinostat, breastfeeding should be discontinued if the mother is treated with belinostat.

Ability to comply with intravenous administration schedule, and the ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the principal investigator.

Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Marked baseline prolongation of Q wave, T wave (QT)/corrected QT(QTc) interval, e.g., repeated demonstration of a QTc interval greater than 500 msec (Fridericia's formula used for correction); Long QT Syndrome. Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes.

Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with belinostat.(HIV) positive patients not receiving antiretroviral therapy are excluded due to the possibility that belinostat may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to belinostat.

Patients may not be receiving any other investigational agents.

History of another invasive malignancy in the last five years. Adequately treated non-invasive, non-melanoma skin cancers as well as in situ carcinoma of the cervix will be allowed.

Prior treatment with drugs of the HDAC inhibitor class.

Patients with tumor amenable to potentially curative therapy as assessed by the investigator.

Subjects with resectable tumors would not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-12; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (2):
- United States (2):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Giaccone G, Wilmink H, Paul MA, van der Valk P. Systemic treatment of malignant thymoma: a decade experience at a single institution. Am J Clin Oncol. 2006 Aug;29(4):336-44. doi: 10.1097/01.coc.0000227481.36109.e7. PMID 16891859
- [Background] Wright CD. Management of thymomas. Crit Rev Oncol Hematol. 2008 Feb;65(2):109-20. doi: 10.1016/j.critrevonc.2007.04.005. Epub 2007 Jun 14. PMID 17570676
- [Background] Giaccone G. Treatment of malignant thymoma. Curr Opin Oncol. 2005 Mar;17(2):140-6. doi: 10.1097/01.cco.0000152628.43867.8e. PMID 15725919
- [Result] Giaccone G, Rajan A, Berman A, Kelly RJ, Szabo E, Lopez-Chavez A, Trepel J, Lee MJ, Cao L, Espinoza-Delgado I, Spittler J, Loehrer PJ Sr. Phase II study of belinostat in patients with recurrent or refractory advanced thymic epithelial tumors. J Clin Oncol. 2011 May 20;29(15):2052-9. doi: 10.1200/JCO.2010.32.4467. Epub 2011 Apr 18. PMID 21502553
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0033.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: United States Food & Drug Administration Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: RECIST — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study plans to accrue 1.85 patients per month. The expected accrual is 41 patients (25 thymoma and 16 thymic).
Period: Overall Study
Arm/Group | Belinostat Treatment
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belinostat Treatment
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.53 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Partial Response
Description: Response is defined by the Response Evaluation Criteria in Solid Tumor (RECIST). Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. For additional details about the RECIST criteria see the protocol Link module.
Time Frame: 25.5 months
Measure: Number; unit: Participants
Groups:
- Thymoma Patients: Well differentiated neoplasm
- Thymic Patients: Poorly differentiated neoplasm
Arm/Group | Thymoma Patients | Thymic Patients
Number analyzed (Participants) | 25 | 16
Participants | 2 [2.3 to 25.9] | 0 [0 to 19.4]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 26 months
Measure: Number; unit: Participants
Groups:
- Belinostat: 1000 mg/m^2 day, 30 minute intravenous infusion daily for 5 days every 3 weeks (day 1-5 of the 3 week treatment cycle). After 12 cycles of treatment, cycles will be given for 5 days every 4 weeks.
Arm/Group | Belinostat
Number analyzed (Participants) | 41
Participants | 41

3. Primary Outcome: Chromosomal Gains or Losses in Comparative Genomic Hydridization in Thymoma and Thymic Cancer
Description: Utilize a patients tumor tissue to determine if there is any correlation between chromosomal gains or losses in comparative genomic hybridization in thymoma and thymic carcinomas and clinical outcomes.
Time Frame: 46 months
Population: Unpublished data from Dr. Giaccone's lab does not reveal an association between these parameters and outcomes in patients with thymic malignancies. Hence we do not plan to perform analyses for these outcome measures and there is no known negative clinical implications associated with this.
Arm/Group | Thymoma Patients | Thymic Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Description: CTCAE v3.0 from beginning of study through 12/31/10; CTCAE v4.0 beginning 1/1/11.
Arm/Group | Belinostat Treatment
Serious Adverse Events (participants affected / at risk) | 6/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belinostat Treatment (N=41)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Infections and infestations-Other, specify infection with normal ANC or Gr 1 or 2 neutrophils:Blood (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belinostat Treatment (N=41)
Anemia (Blood and lymphatic system disorders) | 27 (54)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (8)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Right side abdominal pain
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (14)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 23 (61)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (22)
Chills (General disorders) | 2 (2)
Edema face (General disorders) | 1 (2) — Facial swelling
Edema limbs (General disorders) | 1 (1) — Right lower extremity swelling
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (21)
Fever (General disorders) | 9 (12)
Injection site reaction (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain (General disorders) | 1 (1) — Body aches
Pain (General disorders) | 1 (1) — Head/neck pain
Pain (General disorders) | 1 (1) — Left side
Pain (General disorders) | 1 (2) — Right side pain
Allergic reaction (Immune system disorders) | 8 (10)
Bronchial infection (Infections and infestations) | 1 (2)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations-Other, specify (Infections and infestations) | 1 (1) — HPV (Human papilloma virus)
Lung infection (Infections and infestations) | 1 (1) — Pneumonia
Mucosal infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (5)
Upper respiratory infection (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 2 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 11 (15)
Alanine aminotransferase increased (Investigations) | 8 (10)
Alkaline phosphatase increased (Investigations) | 8 (11)
Blood bilirubin increased (Investigations) | 8 (14)
CPK increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 5 (6)
Electrocardiogram QT corrected interval prolonged (Investigations) | 21 (77)
Lipase increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 20 (92)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (13)
Platelet count decreased (Investigations) | 6 (31)
Serum amylase increased (Investigations) | 1 (2)
Weight gain (Investigations) | 3 (7)
Weight loss (Investigations) | 6 (6)
White blood cell decreased (Investigations) | 14 (33)
Anorexia (Metabolism and nutrition disorders) | 11 (17)
Hypercalcemia (Metabolism and nutrition disorders) | 7 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (17)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 (55)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 5 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (12)
Hyponatremia (Metabolism and nutrition disorders) | 13 (18)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Right chest
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Back spasms
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — L arm
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) — L thigh
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Right arm pain
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — shoulder
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) — Lightheaded
Dizziness (Nervous system disorders) | 4 (7)
Dysgeusia (Nervous system disorders) | 1 (1) — Metallic taste
Dysgeusia (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1) — Slurred speech
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) — L arm
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) — Numb right foot
Peripheral sendory neuropathy (Nervous system disorders) | 1 (1) — Tender skin
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Syncope (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hemoptysis
Bronchopulomonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 9 (11)
Phlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 13 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No